CLINICAL TRIAL: NCT06726473
Title: Validation of the Accuracy of a Novel POCT Dry Blood Gas Analyzer in Acute Care Settings:A Cross-Sectional Study
Brief Title: Validation of the Accuracy of a Novel POCT Dry Blood Gas Analyzer in Acute Care Settings
Status: Completed | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-KY-408-01
Record Dates: First submitted 2024-12-04; First posted 2024-12-10 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Failure; Acid-Base Balance Disorder; Sepsis; Shock; Acute Respiratory Distress Syndrome (ARDS)
Keywords: blood gas analysis; accuracy; EG-i30; Eaglenos
MeSH Terms: conditions — Respiratory Insufficiency; Sepsis; Shock; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Arterial whole blood samples from patients who require blood gas analysis as part of their clinical care will be used. After initial analysis using the ABL90 blood gas analyzer, the remaining samples will be measured with the EG-i30 analyzer for comparison. No DNA will be extracted from these samples, and they will be retained only for the purpose of this study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: ABL90 Group: Blood gas and biochemical measurements are performed using the ABL90 blood gas analyzer. The results will be compared with those from the EG-i30 analyzer.
  Interventions: Diagnostic Test: Wet Blood Gas Analyzer (ABL90)
- Group 2: EG-i30 Group: Blood gas and biochemical measurements are performed using the EG-i30 blood gas analyzer. The results will be compared with those from the ABL90 analyzer.
  Interventions: Diagnostic Test: Dry Blood Gas Analyzer (EG-i30)

INTERVENTIONS:
Diagnostic Test: Wet Blood Gas Analyzer (ABL90) — This group involves the use of the ABL90 wet blood gas analyzer for measuring arterial whole blood samples. The results obtained from the ABL90 analyzer will be compared with those obtained from the EG-i30 dry blood gas analyzer
  Groups: Group 1: ABL90 Group
Diagnostic Test: Dry Blood Gas Analyzer (EG-i30) — This group involves the use of the EG-i30 dry blood gas analyzer for measuring arterial whole blood samples. The results obtained from the EG-i30 analyzer will be compared with those obtained from the ABL90 wet blood gas analyzer.
  Groups: Group 2: EG-i30 Group

SUMMARY:
The goal of this observational study is to validate the performance of the novel POCT dry blood gas analyzer EG-i30, against the currently widely used traditional wet blood gas analyzer, Radiometer ABL90, in acute care settings. The main questions it aims to answer are:

1. How consistent are the results between EG-i30 and ABL90 in acute care settings, including outliers, correlation, linearity, and bias?
2. Whether EG-i30 can be considered a suitable alternative to ABL90 in acute care settings.

Participants will be patients in the emergency department who will undergo simultaneous testing with EG-i30 and ABL90 during their emergency care to assess the performance of EG-i30.

DETAILED DESCRIPTION:
This observational study aims to compare the performance of two blood gas analyzers, the EG-i30 dry blood gas analyzer and the ABL90 wet blood gas analyzer, in an emergency department (ED) or emergency intensive care unit (ICU) setting. The study will evaluate the consistency, correlation, and bias between the two analyzers for various blood gas and biochemical parameters, such as Potential of hydrogen (pH), Partial pressure of oxygen (PaO2), Partial pressure of carbon dioxide (PaCO2), Sodium (Na+), Potassium (K+), Chloride (Cl-), Ionized calcium (iCa2+), Lactate (Lac), Glucose (Glu), and Hematocrit (Hct). The study design is observational, with no intervention or treatment assigned to the participants. The comparison will be made using residual blood samples collected as part of routine care, following standard clinical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo arterial blood gas analysis in the emergency department (ED) or emergency intensive care unit (EICU).

Exclusion Criteria:

* Patients with a confirmed history of infectious diseases such as hepatitis B, syphilis, HIV/AIDS, etc.
* Patients whose residual blood samples are not tested within the specified time frame after collection.
* Other patients deemed ineligible by the investigator (e.g., samples with contamination or other factors affecting sample quality).

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients presenting to the emergency department (ED) or admitted to the emergency intensive care unit (ICU) who are scheduled to undergo arterial blood gas analysis.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Consistency between EG-i30 and ABL90 analyzers for blood gas and biochemical parameters. | Within 2 minutes after arterial blood sample collection
  This outcome measures is to evaluate the consistency between the EG-i30 dry blood gas analyzer and the ABL90 wet blood gas analyzer. Consistency will be assessed by comparing the results of blood gas and biochemical parameters (e.g., pH, PaO2, PaCO2, Na+, K+, Cl-, iCa2+, Lac, Glu, and Hct) and will be evaluated using Bland-Altman analysis.
Correlation between EG-i30 and ABL90 analyzers for blood gas and biochemical parameters. | Within 2 minutes after arterial blood sample collection
  This outcome measures the correlation between the EG-i30 and ABL90 analyzers for blood gas and biochemical parameters (e.g., pH, PaO2, PaCO2, Na+, K+, Cl-, iCa2+, Lac, Glu, and Hct). The correlation will be quantified using Pearson's correlation coefficient.
Bias at clinical decision levels between EG-i30 and ABL90 analyzers. | Within 2 minutes after arterial blood sample collection
  This outcome measure is to evaluate the bias at clinical decision levels between the EG-i30 and ABL90 analyzers. Bias will be assessed by calculating the difference in the results of key blood gas and biochemical parameters (e.g., pH, PaO2, PaCO2, Na+, K+, Cl-, iCa2+, Lac, Glu, and Hct) between the two analyzers at clinically relevant thresholds. These thresholds will be based on established clinical decision points where treatment decisions are made.
Outlier Detection in Blood Gas and Biochemical Parameters | Within 2 minutes after arterial blood sample collection
  This outcome measure aims to identify and evaluate outliers in the blood gas and biochemical parameters (e.g., pH, PaO2, PaCO2, Na+, K+, Cl-, iCa2+, Lac, Glu, and Hct) measured by the EG-i30 and ABL90 analyzers. Outliers will be detected using statistical methods such as the Grubbs test or the Interquartile Range (IQR) method. The impact of these outliers on the consistency and accuracy of the measurements will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Lixia Yang, Principal Investigator — Zhujiang Hospital, Southern Medical University Organization
Locations (1):
- Zhujiang Hospital, Southern Medical University Organization, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Data will be made available to qualified researchers upon submission of a research proposal and execution of a data use agreement. Data access will be granted after the final study results are published and after an ethical review by the institution's ethics board. Data sharing will be coordinated via email. Qualified researchers can contact zjyyllxs@126.com to request access to the data.

REFERENCES:
- [Background] Breathnach CS. The development of blood gas analysis. Med Hist. 1972 Jan;16(1):51-62. doi: 10.1017/s0025727300017257. No abstract available. PMID 4558439
- [Background] Shapiro BA. The history of pH and blood gas analysis. Respir Care Clin N Am. 1995 Sep;1(1):1-5. PMID 9390846
- [Background] Davis MD, Walsh BK, Sittig SE, Restrepo RD. AARC clinical practice guideline: blood gas analysis and hemoximetry: 2013. Respir Care. 2013 Oct;58(10):1694-703. doi: 10.4187/respcare.02786. Epub 2013 Jul 30. PMID 23901131